CLINICAL TRIAL: NCT06129227
Title: Using Functional Near-infrared Spectroscopy to Study the Changes in Brain Activity During Dual-task Walking and the Effects of Structured Cognitive-motor Exercise in Individuals With Stroke
Brief Title: Brain Activity Changes After Structured Cognitive-motor Exercise for People With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Chair professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0037680
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: Dual-task training; Cognitive-motor interference
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: After stratification according to gender and walking speed, the participants will be randomly allocated to one of three groups: (1) dual-task training, (2) single-task training, and (3) control intervention, using a 1:1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: This will be a single-blinded RCT. The assessor will be blinded during assessments. The participants and investigators (trainers) are not possible to be blinded as it is an exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual-task training (Experimental): Mobility tasks performed in conjunction with cognitive tasks
  Interventions: Behavioral: Dual-task training
- Single-task training (Active Comparator): Separate cognitive and mobility exercises
  Interventions: Behavioral: Single-task training
- Control group (Active Comparator): Upper limb strengthening and flexibility exercises
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Dual-task training — This group will receive 30 min of dual-task exercise training and 30 min of stretching exercises in each session. The dual-task component involves walking activities performed in conjunction with cognitive activities. For the stretching exercise component, no cognitive load will be added.
  Arms: Dual-task training
Behavioral: Single-task training — This group will undergo 30 min of single-task mobility training and another 30 min of single-task cognitive activities. The cognitive and mobility exercises will be the same as those in the dual-task group, but they will be performed separately. No extra cognitive load will be imposed during the mobility exercises. No additional motor demand will be imposed during the cognitive exercises, as the participants will be sitting.
  Arms: Single-task training
Behavioral: Control group — This group will undergo 30 min of stretching exercises (same as the dual-task group) and another 30 min of upper limb strengthening exercises performed primarily in the sitting or lying position. No cognitive load will be added.
  Arms: Control group

SUMMARY:
To assess the effects of a dual-task exercise program on cognitive-motor interference during dual-task walking and the associated changes in brain activity.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of chronic disability in Hong Kong and other parts of the world. Mobility dysfunctions are among the most common impairments observed after stroke. Restoration of mobility is also a top priority in rehabilitation goal-setting by stroke patients. In daily life, functional ambulation in the community requires the ability to maintain walking balance while simultaneously engaging in other attention-demanding tasks (i.e., dual-tasking), such as walking when holding a conversation, or crossing the street while attending to traffic signals. There is increasing evidence that performing a cognitive task in conjunction with a mobility task would cause more severe degradation of one or both tasks among stroke patients when compared with age-matched able-bodied individuals. This phenomenon, termed "cognitive-motor interference", should warrant detailed study, since it has an important impact on community-living among people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke confirmed by brain scan reports
* Community-living
* Stroke onset ≥ 6 months
* Aged 50 years or older
* Modified Rankin scale 1-3
* Capable of following verbal instructions
* Montreal Cognitive Assessment score ≥ 22
* Ability to walk for 1 min independently with or without a walking aid
* Not receiving formal rehabilitation elsewhere

Exclusion Criteria:

* Other neurological disorders
* Pain or other comorbidities that seriously affect the ability to walk
* Contraindications to exercise (e.g., angina).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dual-task gait speed | Through study completion, an average of 1 year
  Gait speed under dual-task condition will be recorded
Dual-task cognitive performance | Through study completion, an average of 1 year
  Number of correct responses will be measured during dual-task walking

SECONDARY OUTCOMES:
Dual-task gait performance 1 | Through study completion, an average of 1 year
  Gait cadence will be measured during dual-task walking
Dual-task gait performance 2 | Through study completion, an average of 1 year
  Stride length will be measured during dual-task walking
Dual-task gait performance 3 | Through study completion, an average of 1 year
  Trunk stability will be measured during dual-task walking
Oxyhemoglobin concentration changes of the brain | Through study completion, an average of 1 year
  Oxyhemoglobin concentration changes will be measured using functional near infra-red spectroscopy during dual-task walking

OTHER OUTCOMES:
Single-task walking speed | Through study completion, an average of 1 year
  10-meter walking test will be used to assess single-task walking speed in meters per second
Balance 1 | Through study completion, an average of 1 year
  Mini Balance Evaluation Systems Test will be used to assess postural control, with total points from 0-28. Higher points indicate better performance.
Balance 2 | Through study completion, an average of 1 year
  Activities-specific Balance Confidence Scale will be used to assess confidence of functional balance performance, with total points from 0-100. Higher points indicate better performance.
Cognitive performance | Through study completion, an average of 1 year
  Stroop color word test will be used to assess executive function
Cognitive performance 1 | Through study completion, an average of 1 year
  Digit Span Test will be used to assess working memory
Cognitive performance 2 | Through study completion, an average of 1 year
  Montreal Cognitive Assessment will be used to assess global cognition, with total points from 0-30. Higher points indicate better performance.
Fall incidence | Through study completion, an average of 1 year
  Monthly telephone interviews for recording fall incidence

CONTACTS AND LOCATIONS:
Overall Officials: Marco Yiu Chung PANG, PhD, Principal Investigator — The Hong Kong Polytechnic University; Xun LI, MSc, Study Director — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The study data can be provided via contacting the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From Dec 2025 onwards
Access Criteria: By contacting the Principal Investigator (Prof. Marco PANG): Marco.Pang@polyu.edu.hk